CLINICAL TRIAL: NCT05624424
Title: Effect of Rematazolam Besylate, Propofol, and Sevoflurane Perioperative Sedation on Incidence of Emergence Agitation and Hemodynamics in Patients Undergoing Laparoscopic Abdominal Surgery
Status: Unknown | Phase: Phase 4 | Type: Interventional
Last Known Status: Not yet recruiting
Sponsor: Second Affiliated Hospital of Nanchang University (Other)
Collaborators: Yichang Humanwell Pharmaceutical Co., Ltd., China (Industry)
Responsible Party: Principal Investigator, Fuzhou Hua, Chief Physician, Second Affiliated Hospital of Nanchang University
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Prevention
Other Study IDs: 2022-EA-2
Record Dates: First submitted 2022-11-07; First posted 2022-11-22 (Actual); Last update posted 2022-11-22 (Actual); Status verified 2022-11

CONDITIONS: Emergence Agitation; Remimazolam Besylate; Perioperative Sedation; Laparoscopic Abdominal Surgery; Anesthesia, General
Keywords: Emergence Agitation; Remimazolam Besylate; Propofol; Sevoflurane; Laparoscopic Abdominal Surgery; Perioperative Sedation; Anesthesia, General
MeSH Terms: conditions — Emergence Delirium | interventions — Propofol; Sevoflurane; Sufentanil; cisatracurium; Remifentanil

STUDY DESIGN:
Intervention Model Description: This is a RCTs.
Who Masked: Participant, Outcomes Assessor
Masking Description: Care provider and investigator (anesthesiologist) cannot be blinded for different appearance of remimazolam, propofol and sevoflurane.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (3):
- Remimazolam Besylate (Experimental): Induction of anesthesia Slowly inject Remimazolam Besylate 0.3~0.5 mg/kg (about 1 minute) until loss of consciousness (LoC) and BIS<60, if the degree of sedation is insufficient, additional Remimazolam Besylate (0.05 mg/kg each time) is allowed. After the LoC, sufentanil 0.3~0.5 ug/kg and cisatracurium besilate 0.2-0.3 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  Interventions: Drug: Rematazolam Besylate; Drug: Sufentanil; Drug: Cisatracurium Besylate; Drug: Remifentanil
- Propofol (Active Comparator): Induction of anesthesia Slowly inject Propofol 2~2.5 mg/kg (about 1 minute) until loss of consciousness (LoC) and BIS<60, if the degree of sedation is insufficient, additional Propofol (0.5 mg/kg each time) is allowed. After the LoC, sufentanil 0.3~0.5 ug/kg and cisatracurium besilate 0.2-0.3 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  Interventions: Drug: Propofol; Drug: Sufentanil; Drug: Cisatracurium Besylate; Drug: Remifentanil
- Sevoflurane (Active Comparator): Induction of anesthesia Slowly inject Etomidate 0.03 mg/kg (about 1 minute) until loss of consciousness (LoC) and BIS<60, if the degree of sedation is insufficient, additional etomidate (0.03 mg/kg each time) is allowed. After the LoC, sufentanil 0.3~0.5 ug/kg and cisatracurium besilate 0.2-0.3 mg/kg are injected intravenously. After the muscles are sufficiently relaxed and blood circulation is stable, the tracheal tube is inserted under a glide scope.
  Interventions: Drug: Sevoflurane; Drug: Sufentanil; Drug: Cisatracurium Besylate; Drug: Remifentanil

INTERVENTIONS:
Drug: Rematazolam Besylate — Anesthesia was induced with Rematazolam Besylate 0.3~0.5 mg/kg (about 1 minute) by intravenous injection until the loss of consciousness (LoC) and BIS<60, followed by remimazolam 1-3 mg/kg/h until the end of surgery.
  Arms: Remimazolam Besylate
Drug: Propofol — Anesthesia was induced with Propofol 2~2.5 mg/kg (about 1 minute) by intravenous injection until the loss of consciousness (LoC) and BIS<60, followed by remimazolam 5~12 mg/kg/h until the end of surgery.
  Arms: Propofol
Drug: Sevoflurane — Anesthesia was induced with etomidate 0.03 mg/kg (about 1 minute) by intravenous injection until the loss of consciousness (LoC) and BIS<60, followed by 2 %-3 % Sevoflorane until the end of surgery.
  Arms: Sevoflurane
Drug: Sufentanil — Anesthesia was induced with Sufentanil 0.3~0.5 ug/kg by intravenous injection after the LoC and BIS<60.
Drug: Cisatracurium Besylate — Anesthesia was induced with cisatracurium besilate 0.2-0.3 mg/kg by intravenous injection after the LoC and BIS<60, followed by 0.1 mg/kg/h Cisatracurium Besylate during the operation.
Drug: Remifentanil — After the LoC, remifentanil 0.1~0.3 ug/kg/min inject intravenously until the end of surgery.

SUMMARY:
Emergence agitation (EA) is a transient, self-limited, non-fluctuating state of psychomotor excitement, which closely revolves around the emergence of general anesthesia. Uncontrolled EA during the recovery period increases the potential risk of injury to patients and medical staff, resulting in varying degrees of adverse consequences, such as elevated blood pressure, incision rupture, bleeding, cardio-cerebrovascular accidents and so on, leading to a great waste of resources.

Accumulating scientific evidence indicates that the incidence of EA is related to the use of perioperative sedative drugs. As a novel ultra-short-acting benzodiazepines drugs, Remimazolam has been accepted for induction and maintenance of clinical anesthesia. Compared to traditional benzodiazepines drugs, Remimazolam combines the safety of midazolam with the effectiveness of propofol, and also has the advantages of acting quickly, short half-life, no injection pain, slight respiratory depression, independent of liver and kidney metabolism, long-term infusion without accumulation, and has a specific antagonist: flumazenil. This study aims to investigate whether perioperative sedation of Remimazolam besylate, propofol, and sevoflurane have different effects on the incidence of emergence agitation and hemodynamics in patients undergoing laparoscopic abdominal surgery.

ELIGIBILITY:
Inclusion Criteria:

* 1 Aged 18-65 years, sex was not limited;
* 2 BMI 18-30kg/m2;
* 3 Patients were scheduled for elective laparoscopic abdominal surgery under general anesthesia, the operation time 2h~4h;
* 4 ASA Ⅰ-III;

Exclusion Criteria:

* 1 Relative contraindications to general anesthesia: Patients with severe heart and lung disease, severe infection, uncontrolled hypertension, diabetes, and severe diabetic complications;
* 2 Abnormal renal and liver function: AST or ALT≥2.5×ULN, TBIL≥1.5×ULN, Serum creatinine concentration (SCC)≥1.5×ULN;
* 3 People with a history of mental illness or long-term use of psychotropic drugs (dementia, schizophrenia), chronic analgesic drug use, alcoholism, and cognitive impairment;
* 4 Any cardiovascular or cerebrovascular accidents occurred within 3 months, such as myocardial infarction, stroke, transient ischemic attack;
* 5 Female pregnant patients;
* 6 Patients undergoing hepatobiliary surgery;
* 7 Allergy to the experimental drug;
* 8 Unable to cooperate to complete the test, the patient or family member rejected the participant;

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 1317 (Estimated)
Dates: Start 2022-11-15 (Estimated); Primary Completion 2023-10-31 (Estimated); Study Completion 2023-10-31 (Estimated)

PRIMARY OUTCOMES:
The incidence of emergence agitation | Duration from the time patients awakening to the time of departure from post-anesthesia care unit (PACU), average 1 hour.
  The Riker Sedation-Agitation Scale (RSAS) score ≥ 5 points indicates the presence of emergence agitation.
The incidence of emergence agitation | Duration from the time patients awakening to the time of departure from PACU, average 1 hour.
  The Richmond Agitation-Sedation Scale (RASS) ≥ +1 points indicates the presence of emergence agitation.

SECONDARY OUTCOMES:
Systolic pressure | "30 minutes before intubation", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the post-anesthesia care unit, in about six hours", " mornings and afternoons on the 1st, 3rd and 7th day after operation".
Diastolic pressure | "30 minutes before intubation", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the post-anesthesia care unit, in about six hours", " mornings and afternoons on the 1st, 3rd and 7th day after operation".
Mean pressure | "30 minutes before intubation", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the post-anesthesia care unit, in about six hours", " mornings and afternoons on the 1st, 3rd and 7th day after operation".
Heart rate | "30 minutes before intubation", "immediately after intubation", "every 5 minutes after intubation until the patient leaves the post-anesthesia care unit, in about six hours", " mornings and afternoons on the 1st, 3rd and 7th day after operation".
Recovery times | Duration from the time patients awakening to the time of departure from PACU, average 1 hour.
  Recovery times is defined as the period from discontinuation of anesthetic drugs to the recovery of the patient's self-consciousness and can respond correctly to external stimuli.
Delayed emergence | Duration from the time patients awakening to the time of departure from PACU, average 1 hour.
  Delayed emergence is defined as failure to shake hands and no significant response to nociceptive stimuli more than 30 minutes after surgery.
The incidence of postoperative delirium | Record in the mornings on the 1st, 3rd and 7th day after operation.
  The incidence of postoperative delirium was assessed using CAM Scale.
Postoperative Pain | Record in the mornings on the 1st, 3rd and 7th day after operation.
  The Numericrating scale (NRS) is grouped from 0 to 10. The degree of pain increased directly with the score.
Complication | During the perioperative period, up to 1 week.
  All the perioperative complications are recorded.
Hospitalization time | After the patient is discharged from the hospital, average 1 week.
  The length of hospital stay is recorded.
Hospital expenses | After the patient is discharged from the hospital, average 1 week.
  Hospitalization costs include total hospitalization costs and anesthesia costs.
30-day all-cause mortality | 30 days after surgery
  30-day all-cause mortality is recorded.

CONTACTS AND LOCATIONS:
Locations (6):
- China (6):
  - People's Hospital of Ganzhou, Ganzhou, Jiangxi
  - the First Affiliated Hospital of Gannan Medical College, Gannan Medical College, Ganzhou, Jiangxi
  - The First People's Hospital of JiuJiang, Jiujiang, Jiangxi
  - the Second Affiliated Hospital of Nanchang University, Nanchang University, Nanchang, Jiangxi
  - Tumor Hospital of Jiangxi Province, Nanchang, Jiangxi
  - Shangrao People's Hospital, Shangrao, Jiangxi